CLINICAL TRIAL: NCT06588660
Title: Phase 1b Study of ST-067 (Decoy-Resistant IL-18) With Teclistamab in Multiple Myeloma
Brief Title: ST-067 and Teclistamab for the Treatment of Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to end of funding.
Sponsor: University of Washington (Other)
Collaborators: Simcha Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1123948; NCI-2024-07236 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20589 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ST-067, teclistamab) (Experimental): Patients receive ST-067 SC on days 1, 8, 15 and 22 of cycle 1, on days 8, 15 and 22 of cycle 2, then on days 1 and 15 of subsequent cycles. Patients also receive teclistamab SC on days 1, 3, 5, 15 and 22 of cycle 2 then on days 1, 8, 15, and 22 or days 1 and 15 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the trial and bone marrow aspiration and biopsy during screening and on study.
  Interventions: Biological: Vevoctadekin; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Other: Medical Chart Review; Drug: Teclistamab; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Vevoctadekin — Given SC
  Other Names: Engineered IL-18 Variant ST-067; Engineered Interleukin-18 Variant ST-067; ST 067; ST-067; ST067
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Drug: Teclistamab — Given SC
  Other Names: JNJ 64007957; JNJ-64007957; JNJ64007957; Teclistamab-cqyv; Tecvayli
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection

SUMMARY:
This phase Ib trial tests the safety, side effects and best dose of ST-067 in combination with teclistamab and how well it works in treating patients with multiple myeloma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). ST-067 is an engineered variant of the human cytokine interleukin-18 that may help the immune system kill cancer cells. Teclistamab is a bispecific antibody that can bind to two different antigens at the same time. Teclistamab binds to B-cell maturation antigen (BCMA), a protein found on some B-cells and myeloma cells, and CD3 on T-cells (a type of white blood cell) and may interfere with the ability of cancer cells to grow and spread. Giving ST-067 in combination with teclistamab may be safe, tolerable and/or effective in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of ST-067 in combination with teclistamab followed by a dose-expansion study.

Patients receive ST-067 subcutaneously (SC) on days 1, 8, 15 and 22 of cycle 1, on days 8, 15 and 22 of cycle 2, then on days 1 and 15 of subsequent cycles. Patients also receive teclistamab SC on days 1, 3, 5, 15 and 22 of cycle 2 then on days 1, 8, 15, and 22 or on days 1 and 15 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the trial and bone marrow aspiration and biopsy during screening and on study.

After completion of study treatment, patients are followed every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma, as defined by the presence of at least one International Myeloma Working Group (IMWG) MM-defining event
* Measurable disease as defined by IMWG criteria, requiring one or more of the following:

  * Serum M-protein ≥ 0.5 g/dL
  * Urine M-protein ≥ 200 mg/24h
  * Involved serum free light chain ratio ≥ 10 mg/dL with abnormal kappa/lambda ratio
  * Measurable plasmacytoma, defined as ≥ 1 lesion with cross-sectional diameter ≥ 2 centimeters)
  * Bone marrow plasma cell percentage ≥ 30%
* Eligibility to receive commercial tec per the Food and Drug Administration (FDA) package insert. This requires (1) at least 4 prior lines of therapy including a proteasome inhibitor (PI), immune modulatory imide drug (IMID), and CD38 monoclonal antibody (mAb); and (2) refractoriness, intolerance, or ineligibility (as deemed by the patient's treating physician) to other established therapies known to provide clinical benefit in MM

  * If the FDA package insert for tec is changed to allow for its use in earlier lines of therapy, the above-mentioned stipulations still apply until a protocol modification is approved
* Age ≥ 18 at study screening
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Anticipated survival of > 3 months
* Estimated glomerular filtration rate (eGFR) ≥ 40 mL/min using the Modification of Diet in Renal Disease equation
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) both ≤ 3 x the lab's upper limit of normal (ULN)
* Total bilirubin ≤ 2 x ULN
* Platelets ≥ 25,000/μL at screening (no more than 1 transfusion in the 7-day period leading up to screening labs)
* Hemoglobin ≥ 7 g/dL at screening (no more than 1 transfusion in the 7-day period leading up to screening labs)
* Absolute neutrophil count (ANC) ≥ 1000 cells/mm^3 at screening (no more than one administration of growth factor in the 7-day period leading up to screening labs)
* For patients of reproductive potential only: Willingness to use an effective contraceptive method before, during, and for at least 5 months after the last dose of study therapy
* Ability to understand and provide informed consent as well as willingness to comply with study requirements including visits and biopsies

Exclusion Criteria:

* History of prior BCMA-directed therapy in the past 12 months
* History of another primary malignancy that has not been in remission for at least 1 year

  * However, the following diagnoses are eligible for inclusion: non-melanoma skin cancer, localized prostate cancer, superficial bladder cancer, cervical carcinoma in situ, or any prior malignancy with an estimated > 90% 1-year cure rate per sponsor-investigator
* Any condition requiring systemic treatment with corticosteroids (> 10mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study drug administration. This includes active cytokine release syndrome (CRS), active graft-versus-host disease, or autoimmune conditions

  * Inhaled or topical steroids are allowed, as are replacement corticosteroids for adrenal insufficiency
* Concurrent use of other anti-MM agents or therapies, including investigational drugs, within 7 days of Cycle 1 Day 1

  * Corticosteroids for other purposes, including for pain control, are allowed during the screening period but must also be stopped ≥ 7 days prior to Cycle 1 Day 1
  * Similarly, focal radiation therapy for palliative purposes is permitted during the screening period but must also be completed ≥ 7 days prior to Cycle 1 Day 1
* Known central nervous system (CNS) involvement of MM at time of study screening
* Known active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at time of study screening
* Current pregnancy or breastfeeding, or planned pregnancy or breastfeeding within the next 12 months
* Corrected QT (QTc) interval (Bazett formula) ≥ 500 milliseconds on screening electrocardiogram (ECG)
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Monotherapy dose-limiting toxicities (DLT) rates | Up to 28 days (cycle 1)
  Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) will be graded using American Society for Transplantation and Cellular Therapy (ASTCT) criteria, while other toxicities will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. DLT rates at each dose level will be estimated by isotonic regression by applying the pooled adjacent violators algorithm.
Combination therapy DLT rates | Up to 28 days (cycle 2)
  CRS and ICANS will be graded using ASTCT criteria, while other toxicities will be graded using CTCAE v 5.0. DLT rates at each dose level will be estimated by isotonic regression by applying the pooled adjacent violators algorithm.
Optimal biological dose (OBD) | Up to 28 days
  OBD will be determined based on a composite of clinical information, including safety, tolerability, optimal biological effects without undesirable clinical effects, and biological response data.
Incidence of adverse events (AEs) | Up to 30 days after last dose of ST-067
  The types, frequencies and severity of AEs will be analyzed. CRS and ICANS will be graded using ASTCT criteria, while other toxicities will be graded using CTCAE v 5.0.

SECONDARY OUTCOMES:
Overall response rate (ORR) | At months 1 and 3
  Responses will be assessed per International Myeloma Working Group criteria. ORR will be summarized along with the 2-sided 95% exact Clopper-Pearson confidence interval.
Minimal residual disease (MRD) negativity | At 1 month after initiation of teclistamab
  Bone marrow will be assessed using next generation sequencing for achievement of MRD negativity (threshold 10^-5) and will be compared across all enrolled participants and within each individual.
Duration of response (DOR) | Up to 5 years
  Kaplan-Meier method will be used to analyze DOR.
Progression-free survival (PFS) | From first dose of teclistamab to disease progression or death up to 5 years
  PFS will be calculated using assessments by investigators. Kaplan-Meier methodology will be used to estimate event-free curves and corresponding quartiles (including the median).
Overall survival (OS) | From first dose of teclistamab to death up to 5 years
  Kaplan-Meier methodology will be used to estimate OS curves.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Banerjee, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT06588660/ICF_000.pdf